CLINICAL TRIAL: NCT02117570
Title: A Phase 2, Placebo-controlled, Randomised, Observer-blinded Trial To Evaluate The Safety, Tolerability And Immunogenicity Of A Clostridium Difficile Vaccine Administered As A 3-dose Regimen In Healthy Adults Aged 50 To 85 Years
Brief Title: A Study To Investigate A Clostridium Difficile Vaccine In Healthy Adults Aged 50 to 85 Years, Who Will Each Receive 3 Doses Of Vaccine.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B5091003; 2013-004764-58 (EudraCT Number)
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Results first posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2016-11

CONDITIONS: Clostridium Difficile Associated Disease
Keywords: Clostridium difficile; vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High dose of C. difficile vaccine (Experimental)
  Interventions: Biological: Clostridium difficile vaccine
- Low dose of C. difficile vaccine (Experimental)
  Interventions: Biological: Clostridium difficile vaccine
- Placebo (Placebo Comparator)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Clostridium difficile vaccine — 0.5 mL intramuscular injection on day 1, day 8, and day 30.
  Arms: High dose of C. difficile vaccine
Biological: Clostridium difficile vaccine — 0.5 mL intramuscular injection on day 1, day 8, and day 30.
  Arms: Low dose of C. difficile vaccine
Biological: Placebo — Placebo (0.9 percent saline) given as a 0.5 mL intramuscular injection on day 1, day 8, and day 30.
  Arms: Placebo

SUMMARY:
This study will investigate a Clostridium difficile vaccine in healthy adults aged 50 to 85 years, who will each receive 3 doses of vaccine. The study will assess the safety and tolerability of the vaccine, and also look at the subjects' immune response to the vaccine.

ELIGIBILITY:
Inclusion Criteria:

Healthy male and female subjects aged 50 to 85 years

Exclusion Criteria:

Proven or suspected prior episode of Clostridium difficile associated diarrhea.

Unstable chronic medical condition or disease requiring significant change in therapy or hospitalization for worsening disease within 8 weeks before receipt of study vaccine.

Any contraindication to vaccination or vaccine components, including previous anaphylactic reaction to any vaccine or vaccine-related components.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2014-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- United States (12):
  - Avail Clinical Research, LLC, DeLand, Florida
  - Meridian Clinical Research, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Meridian Clinical Research, Norfolk, Nebraska
  - Meridian Clinical Research, LLC, Omaha, Nebraska
  - Clinical Research Center of Nevada, LLC, Las Vegas, Nevada
  - PMG Research of Charlotte, Charlotte, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - PMG Research of Winston-Salem, Winston-Salem, North Carolina
  - Benchmark Research, Austin, Texas
  - Benchmark Research, San Angelo, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B5091003&StudyName=A%20Phase%202%2C%20Placebo-controlled%2C%20Randomised%2C%20Observer-blinded%20Trial%20To%20Evaluate%20The%20Safety%2C%20Tolerability%20And%20Immunogenicity%20Of%20A%20Clostridium%20Difficile%20Vaccine%20Administered%20As%20A%203-dose%20Regimen%20In%20Healthy%20Adults%20Aged%2050%20To%2085%20Years

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Stage 1, 42 participants aged 50 to 64 years were randomized. After at least 14 days of post-Dose 2 blinded safety data for all Stage 1 participants was reviewed and determined safe, the study proceeded to Stage 2, during which 143 participants aged 65 to 85 years were randomized.
Groups:
- Placebo: Participants were vaccinated with placebo at each vaccination visit (Days 1, 8, and 30) for a total of 3 vaccinations.
- Clostridium Difficile Vaccine, 100 µg: Participants were vaccinated with C difficile vaccine, 100 µg, at each vaccination visit (Days 1, 8, and 30) for a total of 3 vaccinations.
- Clostridium Difficile Vaccine, 200 µg: Participants were vaccinated with C difficile vaccine, 200 µg, at each vaccination visit (Days 1, 8, and 30) for a total of 3 vaccinations.
Period: Stage 1 Participants Aged 50 to 64 Years
Arm/Group | Placebo | Clostridium Difficile Vaccine, 100 µg | Clostridium Difficile Vaccine, 200 µg
Started | 6 (Randomized) | 18 (Randomized) | 18 (Randomized)
Vaccine: Dose 1 | 6 | 18 | 18
Vaccine: Dose 2 | 6 | 18 | 18
Vaccine: Dose 3 | 6 | 17 | 18
Completed | 5 | 15 | 17
Not Completed | 1 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 2 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0
Period: Stage 2 Participants Aged 65 to 85 Years
Arm/Group | Placebo | Clostridium Difficile Vaccine, 100 µg | Clostridium Difficile Vaccine, 200 µg
Started | 21 (Randomized) | 62 (Randomized) | 60 (Randomized)
Vaccine: Dose 1 | 21 | 61 | 60
Vaccine: Dose 2 | 17 | 53 | 50
Vaccine: Dose 3 | 4 | 12 | 12
Completed | 20 | 59 | 54
Not Completed | 1 | 3 | 6
Not completed — Withdrawal by Subject | 0 | 0 | 2
Not completed — Death | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 2 | 2
Not completed — Withdrew before vaccination | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 vaccination
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Clostridium Difficile Vaccine, 100 µg | Clostridium Difficile Vaccine, 200 µg | Total
Number analyzed (Participants) | 27 | 79 | 78 | 184
Age, Customized [Number; unit: Participants]
  Ages 50 to 64 years | 6 | 18 | 18 | 42
  Ages 65 to 85 years | 21 | 61 | 60 | 142
Sex/Gender, Customized [Number; unit: Participants]
  Ages 50 to 64 years: Female | 1 | 5 | 9 | 15
  Ages 50 to 64 years: Male | 5 | 13 | 9 | 27
  Ages 65 to 85 years: Female | 13 | 37 | 36 | 86
  Ages 65 to 85 years: Male | 8 | 24 | 24 | 56

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Prespecified Local Reactions Within 7 Days After Dose 1 (50- to 64-Year Age Cohort)
Description: Pain at injection site: mild=does not interfere with activity; moderate=interferes with activity; severe=prevents daily activity; Grade 4=emergency department visit or hospitalization. Redness/swelling: Mild=2.5 to 5.0 cm; moderate= >5.0 to 10.0 cm; severe= >10 cm; Grade 4=necrosis or exfoliative dermatitis for redness category and only necrosis for swelling category. Any local reaction=any pain at the injection site, any swelling, or any redness.
Time Frame: From Day of Dose 1 vaccination to within 7 days after Dose 1
Population: All randomized participants aged 50 to 64 years who received at least 1 dose of study vaccine
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Clostridium Difficile Vaccine, 100 µg | Clostridium Difficile Vaccine, 200 µg
Number analyzed (Participants) | 6 | 18 | 18
Percentage of participants
  Pain at injection site: Any | 16.7 [0.4 to 64.1] | 16.7 [3.6 to 41.4] | 50.0 [26.0 to 74.0]
  Pain at injection site: Mild | 16.7 [0.4 to 64.1] | 16.7 [3.6 to 41.4] | 50.0 [26.0 to 74.0]
  Pain at injection site: Moderate | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Pain at injection site: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Pain at injection site: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Redness: Any | 0.0 [0.0 to 45.9] | 5.6 [0.1 to 27.3] | 5.6 [0.1 to 27.3]
  Redness: Mild | 0.0 [0.0 to 45.9] | 5.6 [0.1 to 27.3] | 0.0 [0.0 to 18.5]
  Redness: Moderate | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 5.6 [0.1 to 27.3]
  Redness: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Redness: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Swelling: Any | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 16.7 [3.6 to 41.4]
  Swelling: Mild | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 11.1 [1.4 to 34.7]
  Swelling: Moderate | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 5.6 [0.1 to 27.3]
  Swelling: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Swelling: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Any local reaction: Any | 16.7 [0.4 to 64.1] | 16.7 [3.6 to 41.4] | 55.6 [30.78 to 78.5]
  Any local reaction: Mild | 16.7 [0.4 to 64.1] | 16.7 [3.6 to 41.4] | 44.4 [21.5 to 69.2]
  Any local reaction: Moderate | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 11.1 [1.4 to 34.7]
  Any local reaction: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Any local reaction: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]

2. Primary Outcome: Percentage of Participants Reporting Prespecified Local Reactions Within 14 Days After Dose 2 (50- to 64-Year Age Cohort)
Description: as for outcome 1
Time Frame: From Day of Dose 2 vaccination to within 14 days after Dose 2
Population: All randomized participants aged 50 to 64 years who received at least 2 doses of study vaccine
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Clostridium Difficile Vaccine, 100 µg | Clostridium Difficile Vaccine, 200 µg
Number analyzed (Participants) | 6 | 18 | 18
Percentage of participants
  Pain at injection site: Any | 0.0 [0.0 to 45.9] | 61.1 [35.7 to 82.7] | 66.7 [41.0 to 86.7]
  Pain at injection site: Mild | 0.0 [0.0 to 45.9] | 44.4 [21.5 to 69.2] | 55.6 [30.8 to 78.5]
  Pain at injection site: Moderate | 0.0 [0.0 to 45.9] | 16.7 [3.6 to 41.4] | 11.1 [1.4 to 34.7]
  Pain at injection site: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Pain at injection site: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Redness: Any | 16.7 [0.4 to 64.1] | 11.1 [1.4 to 34.7] | 50.0 [26.0 to 74.0]
  Redness: Mild | 16.7 [0.4 to 64.1] | 11.1 [1.4 to 34.7] | 27.8 [9.7 to 53.5]
  Redness: Moderate | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 22.2 [6.4 to 47.6]
  Redness: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Redness: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Swelling: Any | 0.0 [0.0 to 45.9] | 11.1 [1.4 to 34.7] | 27.8 [9.7 to 53.5]
  Swelling: Mild | 0.0 [0.0 to 45.9] | 11.1 [1.4 to 34.7] | 22.2 [6.4 to 47.6]
  Swelling: Moderate | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 5.6 [0.1 to 27.3]
  Swelling: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Swelling: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Any local reaction: Any | 16.7 [0.4 to 64.1] | 61.1 [35.7 to 82.7] | 83.3 [58.6 to 96.4]
  Any local reaction: Mild | 16.7 [0.4 to 64.1] | 44.4 [21.5 to 69.2] | 55.6 [30.8 to 78.5]
  Any local reaction: Moderate | 0.0 [0.0 to 45.9] | 16.7 [3.6 to 41.4] | 27.8 [9.7 to 53.5]
  Any local reaction: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Any local reaction: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]

3. Primary Outcome: Percentage of Participants Reporting Prespecified Local Reactions Within 14 Days After Dose 3 (50- to 64-Year Age Cohort)
Description: as for outcome 1
Time Frame: From Day of Dose 3 vaccination to within 14 days after Dose 3
Population: All randomized participants aged 50 to 64 years who received all 3 doses of study vaccine.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Clostridium Difficile Vaccine, 100 µg | Clostridium Difficile Vaccine, 200 µg
Number analyzed (Participants) | 6 | 17 | 18
Percentage of participants
  Pain at injection site: Any | 0.0 [0.0 to 45.9] | 23.5 [6.8 to 49.9] | 44.4 [21.5 to 69.2]
  Pain at injection site: Mild | 0.0 [0.0 to 45.9] | 23.5 [6.8 to 49.9] | 38.9 [17.3 to 64.3]
  Pain at injection site: Moderate | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 5.6 [0.1 to 27.3]
  Pain at injection site: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  Pain at injection site: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  Redness: Any | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 44.4 [21.5 to 69.2]
  Redness: Mild | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 22.2 [6.4 to 47.6]
  Redness: Moderate | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 22.2 [6.4 to 47.6]
  Redness: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  Redness: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  Swelling: Any | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 33.3 [13.3 to 59.0]
  Swelling: Mild | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 16.7 [3.6 to 41.4]
  Swelling: Moderate | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 16.7 [3.6 to 41.4]
  Swelling: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  Swelling: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  Any local reaction: Any | 0.0 [0.0 to 45.9] | 23.5 [6.8 to 49.9] | 55.6 [30.8 to 78.5]
  Any local reaction: Mild | 0.0 [0.0 to 45.9] | 23.5 [6.8 to 49.9] | 27.8 [9.7 to 53.5]
  Any local reaction: Moderate | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 27.8 [9.7 to 53.5]
  Any local reaction: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  Any local reaction: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]

4. Primary Outcome: Percentage of Participants Reporting Systemic Events Within 7 Days After Dose 1 (50- to 64-Year Age Cohort)
Description: Fever=temperature ≥38.0°C (100.4°C): Mild=38.0°C to 38.4°C (100.4°F-101.1°F); moderate=38.5°C to 38.9°C (101.2°F-102.0°F); severe=39.0°C to 40.0°C (102.1°F-104.0°F); Grade 4= >40.0°C (>104.0°F). Vomiting: Mild=1 to 2 times in 24 hours; moderate= >2 times in 24 hours; severe=requires intravenous hydration; Grade 4=emergency department visit or hospitalization for hypotensive shock. Diarrhea: Mild=2 to 3 loose stools in 24 hours; moderate=4 to 5 loose stools in 24 hours; severe= ≥6 loose stools in 24 hours; Grade 4=emergency department visit or hospitalization. Headache, fatigue, new or worsening joint or muscle pain: Mild=no interference with activity; moderate=some interference with activity; severe=significant interference with activity, prevents daily activity; Grade 4=emergency department visit or hospitalization. Any systemic event: Fever ≥38.0°C, vomiting, diarrhea, headache, fatigue, or new or worsening muscle or joint pain.
Time Frame: From Day of Dose 1 vaccination to within 7 days of Dose 1
Population: All randomized participants aged 50 to 64 years who received at least 1 dose of study vaccine
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Clostridium Difficile Vaccine, 100 µg | Clostridium Difficile Vaccine, 200 µg
Number analyzed (Participants) | 6 | 18 | 18
Percentage of participants
  Fever: Any | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Fever: Mild | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Fever: Moderate | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Fever: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Fever: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Vomiting: Any | 16.7 [0.4 to 64.1] | 5.6 [0.1 to 27.3] | 0.0 [0.0 to 18.5]
  Vomiting: Mild | 16.7 [0.4 to 64.1] | 5.6 [0.1 to 27.3] | 0.0 [0.0 to 18.5]
  Vomiting: Moderate | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Vomiting: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Vomiting: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Diarrhea: Any | 16.7 [0.4 to 64.1] | 22.2 [6.4 to 47.6] | 5.6 [0.1 to 27.3]
  Diarrhea: Mild | 16.7 [0.4 to 64.1] | 22.2 [6.4 to 47.6] | 0.0 [0.0 to 18.5]
  Diarrhea: Moderate | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 5.6 [0.1 to 27.3]
  Diarrhea: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Diarrhea: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Headache: Any | 0.0 [0.0 to 45.9] | 16.7 [3.6 to 41.4] | 5.6 [0.1 to 27.3]
  Headache: Mild | 0.0 [0.0 to 45.9] | 16.7 [3.6 to 41.4] | 0.0 [0.0 to 18.5]
  Headache: Moderate | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 5.6 [0.1 to 27.3]
  Headache: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Headache: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Fatigue: Any | 0.0 [0.0 to 45.9] | 22.2 [6.4 to 47.6] | 11.1 [1.4 to 34.7]
  Fatigue: Mild | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 5.6 [0.1 to 27.3]
  Fatigue: Moderate | 0.0 [0.0 to 45.9] | 22.2 [6.4 to 47.6] | 5.6 [0.1 to 27.3]
  Fatigue: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Fatigue: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  New/worsening muscle pain: Any | 0.0 [0.0 to 45.9] | 11.1 [1.4 to 34.7] | 0.0 [0.0 to 18.5]
  New/worsening muscle pain: Mild | 0.0 [0.0 to 45.9] | 0.0 [0 to 18.5] | 0.0 [0.0 to 18.5]
  New/ worsening muscle pain: Moderate | 0.0 [0.0 to 45.9] | 11.1 [1.4 to 34.7] | 0.0 [0.0 to 18.5]
  New/worsening muscle pain: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  New/worsening muscle pain: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  New/worsening joint pain: Any | 0.0 [0.0 to 45.9] | 11.1 [1.4 to 34.7] | 5.6 [0.1 to 27.3]
  New/worsening joint pain: Mild | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  New/worsening joint pain: Moderate | 0.0 [0.0 to 45.9] | 11.1 [1.4 to 34.7] | 5.6 [0.1 to 27.3]
  New/worsening joint pain: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  New/worsening joint pain: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Any systemic event: Any | 16.7 [0.4 to 64.1] | 44.4 [21.5 to 69.2] | 22.2 [6.4 to 47.6]
  Any systemic event: Mild | 16.7 [0.4 to 64.1] | 22.2 [6.4 to 47.6] | 5.6 [0.1 to 27.3]
  Any systemic event: Moderate | 0.0 [0.0 to 45.9] | 22.2 [6.4 to 47.6] | 16.7 [3.6 to 41.4]
  Any systemic event: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Any systemic event: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]

5. Primary Outcome: Percentage of Participants With A Systemic Event Within 14 Days of Dose 2 (50- to 64-Year Age Cohort)
Description: as for outcome 4
Time Frame: From Day of Dose 2 vaccination to within 14 days after Dose 2
Population: All randomized participants aged 50 to 64 years who received at least 2 doses of study vaccine
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Clostridium Difficile Vaccine, 100 µg | Clostridium Difficile Vaccine, 200 µg
Number analyzed (Participants) | 6 | 18 | 18
Percentage of participants
  Fever: Any | 0.0 [0.0 to 45.9] | 5.6 [0.1 to 27.3] | 5.6 [0.1 to 27.3]
  Fever: Mild | 0.0 [0.0 to 45.9] | 5.6 [0.1 to 27.3] | 5.6 [0.1 to 27.3]
  Fever: Moderate | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Fever: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Fever: Grade 4 | 0.0 [0.0 to 49.5] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Vomiting: Any | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Vomiting: Mild | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Vomiting: Moderate | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Vomiting: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Vomiting: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Diarrhea: Any | 0.0 [0.0 to 45.9] | 11.1 [1.4 to 34.7] | 22.2 [6.4 to 47.6]
  Diarrhea: Mild | 0.0 [0.0 to 45.9] | 5.6 [0.1 to 27.3] | 11.1 [1.4 to 34.7]
  Diarrhea: Moderate | 0.0 [0.0 to 45.9] | 5.6 [0.1 to 27.3] | 11.1 [1.4 to 34.7]
  Diarrhea: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Diarrhea: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Headache: Any | 0.0 [0.0 to 45.9] | 22.2 [6.4 to 47.6] | 33.3 [13.3 to 59.0]
  Headache: Mild | 0.0 [0.0 to 45.9] | 11.1 [1.4 to 34.7] | 22.2 [6.4 to 47.6]
  Headache: Moderate | 0.0 [0.0 to 45.9] | 11.1 [1.4 to 34.7] | 11.1 [1.4 to 34.7]
  Headache: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Headache: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Fatigue: Any | 33.3 [4.3 to 77.7] | 38.9 [17.3 to 64.3] | 33.3 [13.3 to 59.0]
  Fatigue: Mild | 16.7 [0.4 to 64.1] | 16.7 [3.6 to 41.4] | 16.7 [3.6 to 41.4]
  Fatigue: Moderate | 16.7 [0.4 to 64.1] | 16.7 [3.6 to 41.4] | 16.7 [3.6 to 41.4]
  Fatigue: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Fatigue: Grade 4 | 0.0 [0.0 to 45.9] | 5.6 [0.1 to 27.3] | 0.0 [0.0 to 18.5]
  New/worsening muscle pain: Any | 16.7 [0.4 to 64.1] | 27.8 [9.7 to 53.5] | 11.1 [1.4 to 34.7]
  New/worsening muscle pain: Mild | 16.7 [0.4 to 64.1] | 11.1 [1.4 to 34.7] | 5.6 [0.1 to 27.3]
  New/worsening muscle pain: Moderate | 0.0 [0.0 to 45.9] | 16.7 [3.6 to 41.4] | 0.0 [0.0 to 18.5]
  New/worsening muscle pain: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 5.6 [0.1 to 27.3]
  New/worsening muscle pain: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  New/worsening joint pain: Any | 16.7 [0.4 to 64.1] | 33.3 [13.3 to 59.0] | 0.0 [0.0 to 18.5]
  New/worsening joint pain: Mild | 16.7 [0.4 to 64.1] | 27.8 [9.7 to 53.5] | 0.0 [0.0 to 18.5]
  New/worsening joint pain: Moderate | 0.0 [0.0 to 45.9] | 5.6 [0.1 to 27.3] | 0.0 [0.0 to 18.5]
  New/worsening joint pain: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  New/ worsening joint pain: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 0.0 [0.0 to 18.5]
  Any systemic event: Any | 33.3 [4.3 to 77.7] | 44.4 [21.5 to 69.2] | 55.6 [30.8 to 78.5]
  Any systemic event: Mild | 16.7 [0.4 to 64.1] | 16.7 [3.6 to 41.4] | 27.8 [9.7 to 53.5]
  Any systemic event: Moderate | 16.7 [0.4 to 64.1] | 22.2 [6.4 to 47.6] | 22.2 [6.4 to 47.6]
  Any systemic event: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 18.5] | 5.6 [0.1 to 27.3]
  Any systemic event: Grade 4 | 0.0 [0.0 to 45.9] | 5.6 [0.1 to 27.3] | 0.0 [0.0 to 18.5]

6. Primary Outcome: Percentage of Participants Reporting Systemic Events Within 14 Days After Dose 3 (50- to 64-Year Age Cohort)
Description: as for outcome 4
Time Frame: From Day of Dose 3 vaccination to within 14 days after Dose 3
Population: All randomized participants aged 50 to 64 years who received all 3 doses of study vaccine
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Clostridium Difficile Vaccine, 100 µg | Clostridium Difficile Vaccine, 200 µg
Number analyzed (Participants) | 6 | 17 | 18
Percentage of participants
  Fever: Any | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 5.6 [0.1 to 27.3]
  Fever: Mild | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  Fever: Moderate | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  Fever: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 5.6 [0.1 to 27.3]
  Fever: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  Vomiting: Any | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 5.6 [0.1 to 27.3]
  Vomiting: Mild | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 5.6 [0.1 to 27.3]
  Vomiting: Moderate | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  Vomiting: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  Vomiting: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  Diarrhea: Any | 0.0 [0.0 to 45.9] | 41.2 [18.4 to 67.1] | 11.1 [1.4 to 34.7]
  Diarrhea: Mild | 0.0 [0.0 to 45.9] | 29.4 [10.3 to 56.0] | 11.1 [1.4 to 34.7]
  Diarrhea: Moderate | 0.0 [0.0 to 45.9] | 11.8 [1.5 to 36.4] | 0.0 [0.0 to 18.5]
  Diarrhea: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  Diarrhea: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  Headache: Any | 16.7 [0.4 to 64.1] | 29.4 [10.3 to 56.0] | 11.1 [1.4 to 34.7]
  Headache: Mild | 16.7 [0.4 to 64.1] | 23.5 [6.8 to 49.9] | 11.1 [1.4 to 34.7]
  Headache: Moderate | 0.0 [0.0 to 45.9] | 5.9 [0.1 to 28.7] | 0.0 [0.0 to 18.5]
  Headache: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  Headache: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  Fatigue: Any | 33.3 [4.3 to 77.7] | 23.5 [6.8 to 49.9] | 27.8 [9.7 to 53.5]
  Fatigue: Mild | 0.0 [0.0 to 45.9] | 5.9 [0.1 to 28.7] | 16.7 [3.6 to 41.4]
  Fatigue: Moderate | 33.3 [4.3 to 77.7] | 17.6 [3.8 to 43.4] | 11.1 [1.4 to 34.7]
  Fatigue: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  Fatigue: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  New/worsening muscle pain: Any | 16.7 [0.4 to 64.1] | 23.5 [6.8 to 49.9] | 22.2 [6.4 to 47.6]
  New/worsening muscle pain: Mild | 0.0 [0.0 to 45.9] | 17.6 [3.8 to 43.4] | 11.1 [1.4 to 34.7]
  New/worsening muscle pain: Moderate | 16.7 [0.4 to 64.1] | 5.9 [0.1 to 28.7] | 11.1 [1.4 to 34.7]
  New/worsening muscle pain: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  New/worsening muscle pain: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  New/worsening joint pain: Any | 0.0 [0.0 to 45.9] | 23.5 [6.8 to 49.9] | 11.1 [1.4 to 34.7]
  New/worsening joint pain: Mild | 0.0 [0.0 to 45.9] | 11.8 [1.5 to 36.4] | 11.1 [1.4 to 34.7]
  New/worsening joint pain: Moderate | 0.0 [0.0 to 45.9] | 11.8 [1.5 to 36.4] | 0.0 [0.0 to 18.5]
  New/worsening joint pain: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  New/worsening joint pain: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]
  Any systemic event: Any | 33.3 [4.3 to 77.7] | 52.9 [27.8 to 77.0] | 61.1 [35.7 to 82.7]
  Any systemic event: Mild | 0.0 [0.0 to 45.9] | 29.4 [10.3 to 56.0] | 44.4 [21.5 to 69.2]
  Any systemic event: Moderate | 33.3 [4.3 to 77.7] | 23.5 [6.8 to 49.9] | 11.1 [1.4 to 34.7]
  Any systemic event: Severe | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 5.6 [0.1 to 27.3]
  Any systemic event: Grade 4 | 0.0 [0.0 to 45.9] | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 18.5]

7. Primary Outcome: Percentage of Participants Reporting Adverse Events (AEs) to Month 2 and Serious AEs (SAEs) to Month 13 (50- to 64-Year Age Cohort)
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. An SAE is any untoward medical occurrence at any dose that results in death, persistent or significant disability/incapacity, or congenital anomaly/birth defect; is life-threatening; or requires or prolongs inpatient hospitalization.
Time Frame: AEs: From informed consent to Visit 6 (Month 2). SAEs: From informed consent to Visit 9 (Month 13)
Population: All randomized participants aged 50 to 64 years who received at least 1 dose of study vaccine
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | Placebo | Clostridium Difficile Vaccine, 100 µg | Clostridium Difficile Vaccine, 200 µg
Number analyzed (Participants) | 6 | 18 | 18
Participants
  AEs | 16.7 [0.4 to 64.1] | 33.3 [13.3 to 59.0] | 50.0 [26.0 to 74.0]
  SAEs | 16.7 [0.4 to 64.1] | 11.1 [1.4 to 34.7] | 0 [0.0 to 18.5]

8. Primary Outcome: Percentage of Participants With A Local Reaction Within 7 Days of Dose 1 (65- to 85-Year Age Cohort)
Description: as for outcome 1
Time Frame: From Day of Dose 1 vaccination to within 7 days of Dose 1
Population: All randomized participants aged 65 to 85 years who received at least 1 dose of study vaccine.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Clostridium Difficile Vaccine, 100 µg | Clostridium Difficile Vaccine, 200 µg
Number analyzed (Participants) | 21 | 61 | 60
Percentage of participants
  Pain at injection site: Any | 9.5 [1.2 to 30.4] | 24.6 [14.5 to 37.3] | 30.0 [18.8 to 43.2]
  Pain at injection site: Mild | 9.5 [1.2 to 30.4] | 21.3 [11.9 to 33.7] | 28.3 [17.5 to 41.4]
  Pain at injection site: Moderate | 0.0 [0.0 to 16.1] | 3.3 [0.4 to 11.3] | 1.7 [0.0 to 8.9]
  Pain at injection site: Severe | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]
  Pain at injection site: Grade 4 | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]
  Redness: Any | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 6.7 [1.8 to 16.2]
  Redness: Mild | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 3.3 [0.4 to 11.5]
  Redness: Moderate | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 3.3 [0.4 to 11.5]
  Redness: Severe | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]
  Redness: Grade 4 | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]
  Swelling: Any | 0.0 [0.0 to 16.1] | 3.3 [0.4 to 11.3] | 5.0 [1.0 to 13.9]
  Swelling: Mild | 0.0 [0.0 to 16.1] | 1.6 [0.0 to 8.8] | 1.7 [0.0 to 8.9]
  Swelling: Moderate | 0.0 [0.0 to 16.1] | 1.6 [0.0 to 8.8] | 3.3 [0.4 to 11.5]
  Swelling: Severe | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]
  Swelling: Grade 4 | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]
  Any local reaction: Any | 9.5 [1.2 to 30.4] | 27.9 [17.1 to 40.8] | 31.7 [20.3 to 45.0]
  Any local reaction: Mild | 9.5 [1.2 to 30.4] | 23.0 [13.2 to 35.5] | 26.7 [16.1 to 39.7]
  Any local reaction: Moderate | 0.0 [0.0 to 16.1] | 4.9 [1.0 to 13.7] | 5.0 [1.0 to 13.9]
  Any local reaction: Severe | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]
  Any local reaction: Grade 4 | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]

9. Primary Outcome: Percentage of Participants With A Local Reaction Within 14 Days After Dose 2 (65- to 85-Year Age Cohort)
Description: as for outcome 1
Time Frame: From Day of Dose 2 vaccination to 14 days after Dose 2
Population: All randomized participants aged 65 to 85 years who received at least 2 doses of study vaccine
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Clostridium Difficile Vaccine, 100 µg | Clostridium Difficile Vaccine, 200 µg
Number analyzed (Participants) | 17 | 53 | 50
Percentage of participants
  Pain at injection site: Any | 5.9 [0.1 to 28.7] | 66.0 [51.7 to 78.5] | 64.0 [49.2 to 77.1]
  Pain at injection site: Mild | 5.9 [0.1 to 28.7] | 45.3 [31.6 to 59.6] | 48.0 [33.7 to 62.6]
  Pain at injection site: Moderate | 0.0 [0.0 to 19.5] | 18.9 [9.4 to 32.0] | 14.0 [5.8 to 26.7]
  Pain at injection site: Severe | 0.0 [0.0 to 19.5] | 1.9 [0.0 to 10.1] | 2.0 [0.1 to 10.6]
  Pain at injection site: Grade 4 | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 7.1]
  Redness: Any | 0.0 [0.0 to 19.5] | 22.6 [12.3 to 36.2] | 30.0 [17.9 to 44.6]
  Redness: Mild | 0.0 [0.0 to 19.5] | 9.4 [3.1 to 20.7] | 8.0 [2.2 to 19.2]
  Redness: Moderate | 0.0 [0.0 to 19.5] | 5.7 [1.2 to 15.7] | 18.0 [8.6 to 31.4]
  Redness: Severe | 0.0 [0.0 to 19.5] | 7.5 [2.1 to 18.2] | 4.0 [0.5 to 13.7]
  Redness: Grade 4 | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 7.1]
  Swelling: Any | 0.0 [0.0 to 19.5] | 26.4 [15.3 to 40.3] | 26.0 [14.6 to 40.3]
  Swelling: Mild | 0.0 [0.0 to 19.5] | 11.3 [4.3 to 23.0] | 12.0 [4.5 to 24.3]
  Swelling: Moderate | 0.0 [0.0 to 19.5] | 9.4 [3.1 to 20.7] | 12.0 [4.5 to 24.3]
  Swelling: Severe | 0.0 [0.0 to 19.5] | 5.7 [1.2 to 15.7] | 2.0 [0.1 to 10.6]
  Swelling: Grade 4 | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 7.1]
  Any local reaction: Any | 5.9 [0.1 to 28.7] | 67.9 [53.7 to 80.1] | 70.0 [55.4 to 82.1]
  Any local reaction: Mild | 5.9 [0.1 to 28.7] | 34.0 [21.5 to 48.3] | 34.0 [21.2 to 48.8]
  Any local reaction: Moderate | 0.0 [0.0 to 19.5] | 24.5 [13.8 to 38.3] | 30.0 [17.9 to 44.6]
  Any local reaction: Severe | 0.0 [0.0 to 19.5] | 9.4 [3.1 to 20.7] | 6.0 [1.3 to 16.5]
  Any local reaction: Grade 4 | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 7.1]

10. Primary Outcome: Percentage of Participants With A Local Reaction Within 14 Days After Dose 3 (65- to 85-Year Age Cohort)
Description: as for outcome 1
Time Frame: From Day of Dose 3 vaccination to 14 days after Dose 3
Population: All randomized participants aged 65 to 85 years who received all 3 doses of study vaccine
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Clostridium Difficile Vaccine, 100 µg | Clostridium Difficile Vaccine, 200 µg
Number analyzed (Participants) | 4 | 12 | 12
Percentage of participants
  Pain at injection site: Any | 0.0 [0.0 to 60.2] | 25.0 [5.5 to 57.2] | 25.0 [5.5 to 57.2]
  Pain at injection site: Mild | 0.0 [0.0 to 60.2] | 16.7 [2.1 to 48.4] | 16.7 [2.1 to 48.4]
  Pain at injection site: Moderate | 0.0 [0.0 to 600.2] | 8.3 [0.2 to 38.5] | 8.3 [0.2 to 38.5]
  Pain at injection site: Severe | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Pain at injection site: Grade 4 | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Redness: Any | 0.0 [0.0 to 60.2] | 8.3 [0.2 to 38.5] | 8.3 [0.2 to 38.5]
  Redness: Mild | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 8.3 [0.2 to 38.5]
  Redness: Moderate | 0.0 [0.0 to 60.2] | 8.3 [0.2 to 38.5] | 0.0 [0.0 to 26.5]
  Redness: Severe | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Redness: Grade 4 | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Swelling: Any | 0.0 [0.0 to 60.2] | 25.0 [5.5 to 57.2] | 16.7 [2.1 to 48.4]
  Swelling: Mild | 0.0 [0.0 to 60.2] | 16.7 [2.1 to 48.4] | 16.7 [2.1 to 48.4]
  Swelling: Moderate | 0.0 [0.0 to 60.2] | 8.3 [0.2 to 38.5] | 0.0 [0.0 to 26.5]
  Swelling: Severe | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Swelling: Grade 4 | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Any local reaction: Any | 0.0 [0.0 to 60.2] | 33.3 [9.9 to 65.1] | 25.0 [5.5 to 57.2]
  Any local reaction: Mild | 0.0 [0.0 to 60.2] | 16.7 [2.1 to 48.4] | 16.7 [2.1 to 48.4]
  Any local reaction: Moderate | 0.0 [0.0 to 60.2] | 16.7 [2.1 to 48.4] | 8.3 [0.2 to 38.5]
  Any local reaction: Severe | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Any local reaction: Grade 4 | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]

11. Primary Outcome: Percentage of Participants With A Systemic Event Within 7 Days of Dose 1 (65- to 85-Year Age Cohort)
Description: as for outcome 4
Time Frame: From Day of Dose 1 vaccination to within 7 days of Dose 1
Population: All randomized participants aged 65 to 85 years who received at least 1 dose of study vaccine
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Clostridium Difficile Vaccine, 100 µg | Clostridium Difficile Vaccine, 200 µg
Number analyzed (Participants) | 21 | 61 | 60
Percentage of participants
  Fever: Any | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 3.3 [0.4 to 11.5]
  Fever: Mild | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 1.7 [0.0 to 8.9]
  Fever: Moderate | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 1.7 [0.0 to 8.9]
  Fever: Severe | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]
  Fever: Grade 4 | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]
  Vomiting: Any | 0.0 [0.0 to 16.1] | 1.6 [0.0 to 8.8] | 0.0 [0.0 to 6.0]
  Vomiting: Mild | 0.0 [0.0 to 16.1] | 1.6 [0.0 to 8.8] | 0.0 [0.0 to 6.0]
  Vomiting: Moderate | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]
  Vomiting: Severe | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]
  Vomiting: Grade 4 | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]
  Diarrhea: Any | 4.8 [0.1 to 23.8] | 11.5 [4.7 to 22.2] | 15.0 [7.1 to 26.6]
  Diarrhea: Mild | 4.8 [0.1 to 23.8] | 8.2 [2.7 to 18.1] | 11.7 [4.8 to 22.6]
  Diarrhea: Moderate | 0.0 [0.0 to 16.1] | 3.3 [0.4 to 11.3] | 3.3 [0.4 to 11.5]
  Diarrhea: Severe | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]
  Diarrhea: Grade 4 | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]
  Headache: Any | 9.5 [1.2 to 30.4] | 13.1 [5.8 to 24.2] | 15.0 [7.1 to 26.6]
  Headache: Mild | 0.0 [0.0 to 16.1] | 13.1 [5.8 to 24.2] | 8.3 [2.8 to 18.4]
  Headache: Moderate | 9.5 [1.2 to 30.4] | 0.0 [0.0 to 5.9] | 6.7 [1.8 to 16.2]
  Headache: Severe | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]
  Headache: Grade 4 | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]
  Fatigue: Any | 19.0 [5.4 to 41.9] | 26.2 [15.8 to 39.1] | 26.7 [16.1 to 39.7]
  Fatigue: Mild | 14.3 [3.0 to 36.3] | 18.0 [9.4 to 30.0] | 13.3 [5.9 to 24.6]
  Fatigue: Moderate | 4.8 [0.1 to 23.8] | 8.2 [2.7 to 18.1] | 13.3 [5.9 to 24.6]
  Fatigue: Severe | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]
  Fatigue: Grade 4 | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]
  New/worsening muscle pain: Any | 19.0 [5.4 to 41.9] | 4.9 [1.0 to 13.7] | 8.3 [2.8 to 18.4]
  New/worsening muscle pain: Mild | 4.8 [0.1 to 23.8] | 3.3 [0.4 to 11.3] | 6.7 [1.8 to 16.2]
  New/worsening muscle pain: Moderate | 14.3 [3.0 to 36.3] | 1.6 [0.0 to 8.8] | 0.0 [0.0 to 6.0]
  New/worsening muscle pain: Severe | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 1.7 [0.0 to 8.9]
  New/worsening muscle pain: Grade 4 | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]
  New/worsening joint pain: Any | 4.8 [0.1 to 23.8] | 8.2 [2.7 to 18.1] | 8.3 [2.8 to 18.4]
  New/worsening joint pain: Mild | 4.8 [0.1 to 23.8] | 1.6 [0.0 to 8.8] | 5.0 [1.0 to 13.9]
  New/worsening joint pain: Moderate | 0.0 [0.0 to 16.1] | 6.6 [1.8 to 15.9] | 3.3 [0.4 to 11.5]
  New/worsening joint pain: Severe | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]
  New/worsening joint pain: Grade 4 | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]
  Any systemic event: Any | 23.8 [8.2 to 47.2] | 32.8 [21.3 to 46.0] | 45.0 [32.1 to 58.4]
  Any systemic event: Mild | 4.8 [0.1 to 23.8] | 21.3 [11.9 to 33.7] | 23.3 [13.4 to 36.0]
  Any systemic event: Moderate | 19.0 [5.4 to 41.9] | 11.5 [4.7 to 22.2] | 20.0 [10.8 to 32.3]
  Any systemic event: Severe | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 1.7 [0.0 to 8.9]
  Any systemic event: Grade 4 | 0.0 [0.0 to 16.1] | 0.0 [0.0 to 5.9] | 0.0 [0.0 to 6.0]

12. Primary Outcome: Percentage of Participants With a Systemic Event Within 14 Days of Dose 2 (65- to 85-Year Age Cohort)
Description: as for outcome 4
Time Frame: From Day of Dose 2 vaccination to within 14 days after Dose 2
Population: All randomized participants aged 65 to 85 years who received at least 2 doses of study vaccine
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Clostridium Difficile Vaccine, 100 µg | Clostridium Difficile Vaccine, 200 µg
Number analyzed (Participants) | 17 | 53 | 50
Percentage of participants
  Fever: Any | 0.0 [0.0 to 19.5] | 1.9 [0.0 to 10.1] | 4.0 [0.5 to 13.7]
  Fever: Mild | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 6.7] | 2.0 [0.1 to 10.6]
  Fever: Moderate | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 7.1]
  Fever: Severe | 0.0 [0.0 to 19.5] | 1.9 [0.0 to 10.1] | 2.0 [0.1 to 10.6]
  Fever: Grade 4 | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 7.1]
  Vomiting: Any | 0.0 [0.0 to 19.5] | 1.9 [0.0 to 10.1] | 2.0 [0.1 to 10.6]
  Vomiting: Mild | 0.0 [0.0 to 19.5] | 1.9 [0.0 to 10.1] | 0.0 [0.0 to 7.1]
  Vomiting: Moderate | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 6.7] | 2.0 [0.1 to 10.6]
  Vomiting: Severe | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 7.1]
  Vomiting: Grade 4 | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 7.1]
  Diarrhea: Any | 23.5 [6.8 to 49.9] | 17.0 [8.1 to 29.8] | 18.0 [8.6 to 31.4]
  Diarrhea: Mild | 5.9 [0.1 to 28.7] | 7.5 [2.1 to 18.2] | 16.0 [7.2 to 29.1]
  Diarrhea: Moderate | 17.6 [3.8 to 43.4] | 9.4 [3.1 to 20.7] | 0.0 [0.0 to 7.1]
  Diarrhea: Severe | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 6.7] | 2.0 [0.1 to 10.6]
  Diarrhea: Grade 4 | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 7.1]
  Headache: Any | 23.5 [6.8 to 49.9] | 26.4 [15.3 to 40.3] | 14.0 [5.8 to 26.7]
  Headache: Mild | 17.6 [3.8 to 43.4] | 17.0 [8.1 to 29.8] | 12.0 [4.5 to 24.3]
  Headache: Moderate | 5.9 [0.1 to 28.7] | 9.4 [3.1 to 20.7] | 2.0 [0.1 to 10.6]
  Headache: Severe | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 7.1]
  Headache: Grade 4 | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 7.1]
  Fatigue: Any | 17.6 [3.8 to 43.4] | 39.6 [26.5 to 54.0] | 32.0 [19.5 to 46.7]
  Fatigue: Mild | 11.8 [1.5 to 36.4] | 20.8 [10.8 to 34.1] | 20.0 [10.0 to 33.7]
  Fatigue: Moderate | 5.9 [0.1 to 28.7] | 18.9 [9.4 to 32.0] | 12.0 [4.5 to 24.3]
  Fatigue: Severe | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 7.1]
  Fatigue: Grade 4 | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 7.1]
  New/worsening muscle pain: Any | 11.8 [1.5 to 36.4] | 26.4 [15.3 to 40.3] | 24.0 [13.1 to 38.2]
  New/worsening muscle pain: Mild | 0.0 [0.0 to 19.5] | 17.0 [8.1 to 29.8] | 14.0 [5.8 to 26.7]
  New/worsening muscle pain: Moderate | 11.8 [1.5 to 36.4] | 9.4 [3.1 to 20.7] | 10.0 [3.3 to 21.8]
  New/worsening muscle pain: Severe | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 7.1]
  New/worsening muscle pain: Grade 4 | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 7.1]
  New/worsening joint pain: Any | 11.8 [1.5 to 36.4] | 20.8 [10.8 to 34.1] | 14.0 [5.8 to 26.7]
  New/worsening joint pain: Mild | 0.0 [0.0 to 19.5] | 13.2 [5.5 to 25.3] | 10.0 [3.3 to 21.8]
  New/worsening joint pain: Moderate | 11.8 [1.5 to 36.4] | 7.5 [2.1 to 18.2] | 4.0 [0.5 to 13.7]
  New/worsening joint pain: Severe | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 7.1]
  New/worsening joint pain: Grade 4 | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 7.1]
  Any systemic event: Any | 35.3 [14.2 to 61.7] | 50.9 [36.8 to 64.9] | 58.0 [43.2 to 71.8]
  Any systemic event: Mild | 5.9 [0.1 to 28.7] | 17.0 [8.1 to 29.8] | 34.0 [21.2 to 48.8]
  Any systemic event: Moderate | 29.4 [10.3 to 56.0] | 32.1 [19.9 to 46.3] | 20.0 [10.0 to 33.7]
  Any systemic event: Severe | 0.0 [0.0 to 19.5] | 1.9 [0.0 to 10.1] | 4.0 [0.5 to 13.7]
  Any systemic event: Grade 4 | 0.0 [0.0 to 19.5] | 0.0 [0.0 to 6.7] | 0.0 [0.0 to 7.1]

13. Primary Outcome: Percentage of Participants Reporting Systemic Events Within 14 Days After Dose 3 (65- to 85-Year Age Cohort)
Description: as for outcome 4
Time Frame: From Day of Dose 3 vaccination to within 14 days after Dose 3
Population: All randomized participants aged 65 to 85 years who received all 3 doses of study vaccine
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Clostridium Difficile Vaccine, 100 µg | Clostridium Difficile Vaccine, 200 µg
Number analyzed (Participants) | 4 | 12 | 12
Percentage of participants
  Fever: Any | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Fever: Mild | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Fever: Moderate | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Fever: Severe | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Fever: Grade 4 | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Vomiting: Any | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Vomiting: Mild | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Vomiting: Moderate | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Vomiting: Severe | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Vomiting: Grade 4 | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Diarrhea: Any | 25.0 [0.6 to 80.6] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Diarrhea: Mild | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Diarrhea: Moderate | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Diarrhea: Severe | 25.0 [0.6 to 80.6] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Diarrhea: Grade 4 | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Headache: Any | 25.0 [0.6 to 80.6] | 8.3 [0.2 to 38.5] | 8.3 [0.2 to 38.5]
  Headache: Mild | 25.0 [0.6 to 80.6] | 0.0 [0.0 to 26.5] | 8.3 [0.2 to 38.5]
  Headache: Moderate | 0.0 [0.0 to 60.2] | 8.3 [0.2 to 38.5] | 0.0 [0.0 to 26.5]
  Headache: Severe | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Headache: Grade 4 | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Fatigue: Any | 0.0 [0.0 to 60.2] | 33.3 [9.9 to 65.1] | 8.3 [0.2 to 38.5]
  Fatigue: Mild | 0.0 [0.0 to 60.2] | 25.0 [5.5 to 57.2] | 8.3 [0.2 to 38.5]
  Fatigue: Moderate | 0.0 [0.0 to 60.2] | 8.3 [0.2 to 38.5] | 0.0 [0.0 to 26.5]
  Fatigue: Severe | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Fatigue: Grade 4 | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  New/worsening muscle pain: Any | 0.0 [0.0 to 60.2] | 16.7 [2.1 to 48.4] | 0.0 [0.0 to 26.5]
  New/worsening muscle pain: Mild | 0.0 [0.0 to 60.2] | 8.3 [0.2 to 38.5] | 0.0 [0.0 to 26.5]
  New/worsening muscle pain: Moderate | 0.0 [0.0 to 60.2] | 8.3 [0.2 to 38.5] | 0.0 [0.0 to 26.5]
  New/worsening muscle pain: Severe | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  New/worsening muscle pain: Grade 4 | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  New/worsening joint pain: Any | 0.0 [0.0 to 60.2] | 25.0 [5.5 to 57.2] | 0.0 [0.0 to 26.5]
  New/worsening joint pain: Mild | 0.0 [0.0 to 60.2] | 8.3 [0.2 to 38.5] | 0.0 [0.0 to 26.5]
  New/worsening joint pain: Moderate | 0.0 [0.0 to 60.2] | 16.7 [2.1 to 48.4] | 0.0 [0.0 to 26.5]
  New/worsening joint pain: Severe | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  New/worsening joint pain: Grade 4 | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Any systemic event: Any | 50.0 [6.8 to 93.2] | 50.0 [21.1 to 78.9] | 8.3 [0.2 to 38.5]
  Any systemic event: Mild | 25.0 [0.6 to 80.6] | 25.0 [5.5 to 57.2] | 8.3 [0.2 to 38.5]
  Any systemic event: Moderate | 0.0 [0.0 to 60.2] | 25.0 [5.5 to 57.2] | 0.0 [0.0 to 26.5]
  Any systemic event: Severe | 25.0 [0.6 to 80.6] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]
  Any systemic event: Grade 4 | 0.0 [0.0 to 60.2] | 0.0 [0.0 to 26.5] | 0.0 [0.0 to 26.5]

14. Primary Outcome: Percentage of Participants Reporting Adverse Events (AEs) to Month 2 and Serious AEs (SAEs) to Month 13 (65- to 85-Year Age Cohort)
Description: as for outcome 7
Time Frame: AEs: From informed consent to Visit 6 (Month 2). SAEs: From informed consent to Visit 9 (Month 13)
Population: All randomized participants aged 65 to 85 who received at least 1 dose of study vaccine
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Placebo | Clostridium Difficile Vaccine, 100 µg | Clostridium Difficile Vaccine, 200 µg
Number analyzed (Participants) | 21 | 61 | 60
Percentage of participants
  AEs | 38.1 [18.1 to 61.6] | 36.1 [24.2 to 49.4] | 41.7 [29.1 to 55.1]
  SAEs | 14.3 [3.0 to 36.3] | 3.3 [0.4 to 11.3] | 10.0 [3.8 to 20.5]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were assessed from informed consent through and including Visit 6 (Month 2). Serious AEs (SAEs) were assessed from informed consent through and including Visit 9.
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Groups:
- Placebo (50-64 Year Age Cohort); Placebo (65-85 Year Age Cohort): Participants were vaccinated with placebo at each vaccination visit (Days 1, 8, and 30) for a total of 3 vaccinations.
- Clostridium Difficile Vaccine, 100 µg (50-64 Year Age Cohort); Clostridium Difficile Vaccine, 100 µg (65-85 Year Age Cohort): Participants were vaccinated with C difficile vaccine, 100 µg, at each vaccination visit (Days 1, 8, and 30) for a total of 3 vaccinations.
- Clostridium Difficile Vaccine, 200 µg (50-64 Year Age Cohort); Clostridium Difficile Vaccine, 200 µg (65-85 Year Age Cohort): Participants were vaccinated with C difficile vaccine, 200 µg, at each vaccination visit (Days 1, 8, and 30) for a total of 3 vaccinations.
Arm/Group | Placebo (50-64 Year Age Cohort) | Clostridium Difficile Vaccine, 100 µg (50-64 Year Age Cohort) | Clostridium Difficile Vaccine, 200 µg (50-64 Year Age Cohort) | Placebo (65-85 Year Age Cohort) | Clostridium Difficile Vaccine, 100 µg (65-85 Year Age Cohort) | Clostridium Difficile Vaccine, 200 µg (65-85 Year Age Cohort)
Serious Adverse Events (participants affected / at risk) | 1/6 | 2/18 | 0/18 | 3/21 | 2/61 | 6/60
Other Adverse Events (participants affected / at risk) | 0/6 | 5/18 | 9/18 | 5/21 | 22/61 | 22/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (50-64 Year Age Cohort) (N=6) | Clostridium Difficile Vaccine, 100 µg (50-64 Year Age Cohort) (N=18) | Clostridium Difficile Vaccine, 200 µg (50-64 Year Age Cohort) (N=18) | Placebo (65-85 Year Age Cohort) (N=21) | Clostridium Difficile Vaccine, 100 µg (65-85 Year Age Cohort) (N=61) | Clostridium Difficile Vaccine, 200 µg (65-85 Year Age Cohort) (N=60)
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gangrene (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Osteomyelitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pelvic abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Device breakage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Device malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (50-64 Year Age Cohort) (N=6) | Clostridium Difficile Vaccine, 100 µg (50-64 Year Age Cohort) (N=18) | Clostridium Difficile Vaccine, 200 µg (50-64 Year Age Cohort) (N=18) | Placebo (65-85 Year Age Cohort) (N=21) | Clostridium Difficile Vaccine, 100 µg (65-85 Year Age Cohort) (N=61) | Clostridium Difficile Vaccine, 200 µg (65-85 Year Age Cohort) (N=60)
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 1
Injection site erythema (General disorders) | 0 | 1 | 3 | 0 | 2 | 5
Injection site pruritus (General disorders) | 0 | 0 | 1 | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site bruising (General disorders) | 0 | 0 | 0 | 0 | 2 | 0
Injection site induration (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 2
Injection site rash (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pelvic abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Skin candida (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 2 | 2
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Device malfunction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Sinus operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 3
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.